CLINICAL TRIAL: NCT00247676
Title: An Open Label International Multi-Center Phase 2 Activity And Safety Study Of SU011248 In Patients With Unresectable Hepatocellular Carcinoma
Brief Title: An International Phase 2 Study Of SU011248 In Patients With Inoperable Liver Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A6181055
Record Dates: First submitted 2005-11-01; First posted 2005-11-02 (Estimated); Results first posted 2010-02-02 (Estimated); Last update posted 2010-02-18 (Estimated); Status verified 2010-02

CONDITIONS: Liver Neoplasms; Unresectable Hepatocellular Carcinoma
Keywords: Liver neoplasms, sunitinib, Phase 2
MeSH Terms: conditions — Liver Neoplasms | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: Sunitinib (SU011248)

INTERVENTIONS:
Drug: Sunitinib (SU011248) — Sunitinib 50 mg by oral capsule, daily for 4 weeks in every 6 week cycle until progression or unacceptable toxicity.
  Other Names: SU011248, Sutent

SUMMARY:
The study will consist of two parts. In Part 1 the study will start enrolling 38 patients and then further 25 patients up to a total of 63 eligible patients. If the study gives good results it can be expanded to a total of 160 patients. SU011248 will be administered orally daily for 4 weeks followed by a 2-week rest at a starting dose of 50 mg [milligrams] with provision for dose reduction based on tolerability. All patients will receive repeated cycles of SU011248 until disease progression, occurrence of unacceptable toxicity, or other withdrawal criteria are met. After discontinuation of treatment, patients will be followed up in order to collect information on further antineoplastic therapy and survival

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of hepatocellular carcinoma
* Patients must present with disease not amenable to curative surgery (i.e. either hepatectomy, or liver transplant).
* Evidence of measurable disease by radiographic technique
* Adequate organ function.

Exclusion Criteria:

* Prior treatment with any systemic treatment for liver cancer
* Presence of clinically relevant ascites
* Severe hemorrhage <4 weeks of starting study treatment.
* Diagnosis of second malignancy within last 3 years
* History of or known brain metastases, spinal cord compression, or carcinomatous meningitis
* Known human immunodeficiency virus (HIV)
* Serious acute or chronic illness
* Current treatment on another clinical trial
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2006-02; Primary Completion 2008-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- France (3):
  - Pfizer Investigational Site, Clichy
  - Pfizer Investigational Site, Rennes
  - Pfizer Investigational Site, Saint Herrblain Cedex
- Pfizer Investigational Site, Seoul, South Korea
- Pfizer Investigational Site, Taipei, Taiwan

REFERENCES:
- [Derived] Harmon CS, DePrimo SE, Raymond E, Cheng AL, Boucher E, Douillard JY, Lim HY, Kim JS, Lechuga MJ, Lanzalone S, Lin X, Faivre S. Mechanism-related circulating proteins as biomarkers for clinical outcome in patients with unresectable hepatocellular carcinoma receiving sunitinib. J Transl Med. 2011 Jul 25;9:120. doi: 10.1186/1479-5876-9-120. PMID 21787417
- [Derived] Faivre S, Zappa M, Vilgrain V, Boucher E, Douillard JY, Lim HY, Kim JS, Im SA, Kang YK, Bouattour M, Dokmak S, Dreyer C, Sablin MP, Serrate C, Cheng AL, Lanzalone S, Lin X, Lechuga MJ, Raymond E. Changes in tumor density in patients with advanced hepatocellular carcinoma treated with sunitinib. Clin Cancer Res. 2011 Jul 1;17(13):4504-12. doi: 10.1158/1078-0432.CCR-10-1708. Epub 2011 Apr 29. PMID 21531821
- [Derived] Faivre S, Raymond E, Boucher E, Douillard J, Lim HY, Kim JS, Zappa M, Lanzalone S, Lin X, Deprimo S, Harmon C, Ruiz-Garcia A, Lechuga MJ, Cheng AL. Safety and efficacy of sunitinib in patients with advanced hepatocellular carcinoma: an open-label, multicentre, phase II study. Lancet Oncol. 2009 Aug;10(8):794-800. doi: 10.1016/S1470-2045(09)70171-8. Epub 2009 Jul 6. PMID 19586800
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181055&StudyName=An%20International%20Phase%202%20Study%20Of%20SU011248%20In%20Patients%20With%20Inoperable%20Liver%20Cancer

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was designed using a Simon 2-stage design with the objective response rate as the primary efficacy endpoint. Enrollment was halted after the first stage because the minimum number of responders by Response Evaluation Criteria in Solid Tumors (RECIST) needed to continue into Stage 2 was not reached.
Groups:
- 50 Milligram (mg) Sunitinib: Subjects received open-label sunitinib malate at a starting dose of 50 mg once daily for 4 consecutive weeks followed by a 2-week rest period to form a complete cycle of 6 weeks.
Period: Overall Study
Arm/Group | 50 Milligram (mg) Sunitinib
Started | 37
Completed | 1
Not Completed | 36
Not completed — Death | 5
Not completed — Adverse Event | 11
Not completed — Lack of Efficacy | 15
Not completed — Other | 3
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | 50 Milligram (mg) Sunitinib
Number analyzed (Participants) | 37
Age Continuous [Mean (Standard Deviation); unit: years] | 59.0 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 34

OUTCOME MEASURES:

1. Secondary Outcome: Duration of Objective Response (CR or PR)
Description: Time from the first documentation of objective tumor response (CR or PR) that was subsequently confirmed to the first documentation of disease progression or to death due to any cause. CR=disappearance of all target lesions. PR= ≥30% decrease in sum of longest dimensions of lesions taking as reference baseline sum longest dimensions.
Time Frame: From start of treatment until Day 28 of Cycle 1, Day 28 of Cycles thereafter or death due to cancer
Population: From the Overall ITT population, only 1 subject had Objective Response for evaluation of duration of objective response.
Measure: Number; unit: Weeks
Arm/Group | 50 Milligram (mg) Sunitinib
Number analyzed (Participants) | 1
Weeks | 32.4

2. Primary Outcome: Best Overall Response
Description: Number of subjects with best overall response. Complete response (CR)=disappearance of all target lesions. Partial Response (PR)= ≥30% decrease in sum of longest dimensions of lesions taking as reference baseline sum longest dimensions. Progressive disease (PD)= ≥ 20% increase in sum of longest dimensions of lesions taking as a reference smallest sum of the longest dimensions since treatment start, or the appearance of ≥ 1 new lesion. Stable disease (SD)=neither shrinkage for PR or increase for PD taking as reference smallest sum of longest dimensions since treatment start.
Time Frame: From start of treatment until Day 28 of Cycle 1, Day 28 of Cycles thereafter
Population: Intent-to-treat (ITT) population includes all patients enrolled in the study that received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | 50 Milligram (mg) Sunitinib
Number analyzed (Participants) | 37
participants
  CR | 0
  PR | 1
  SD | 15
  Progressive Disease | 11
  Not Evaluable | 7
  Missing | 3

3. Secondary Outcome: Clinical Benefit Response (CR, PR, or SD With Duration ≥12 Weeks)
Description: Number of patients with Clinical Benefit Response: confirmed CR, confirmed PR, or SD for at least 12 weeks on study according to RECIST. CR=disappearance of all target lesions. PR= ≥30% decrease in sum of longest dimensions of lesions taking as reference baseline sum longest dimensions. SD=neither shrinkage for PR or increase for PD taking as reference smallest sum of longest dimensions since treatment start.
Time Frame: From start of treatment until Day 28 of Cycle 1, Day 28 of Cycles thereafter or SD with duration of at least 12 weeks on study
Population: ITT
Measure: Number; unit: participants
Arm/Group | 50 Milligram (mg) Sunitinib
Number analyzed (Participants) | 37
participants | 14
Statistical Analysis 1: Comparison: 50 Milligram (mg) Sunitinib; Test type: Superiority or Other; clinical benefit response rate = 37.8, 95% CI [22.5 to 55.2] — Clinical benefit response rate: percent of patients with confirmed CR, confirmed PR, or SD for at least 12 weeks according to RECIST, relative to total treated patients

4. Secondary Outcome: Best Overall Response of PR or SD With Duration ≥12 Weeks
Description: Number of patients with best overall response of PR or SD with duration ≥ 12 weeks. Best overall response was defined as the time from the first documentation of tumor response that was subsequently confirmed to the first documentation of disease progression or to death due to any cause. CR=disappearance of all target lesions. PR= ≥30% decrease in sum of longest dimensions of lesions taking as reference baseline sum longest dimensions. SD=neither shrinkage for PR or increase for PD taking as reference smallest sum of longest dimensions since treatment start.
Time Frame: From start of treatment until Day 28 of Cycle 1, Day 28 of Cycles thereafter or SD with duration of at least 12 weeks or death due to cancer
Population: ITT
Measure: Number; unit: participants
Arm/Group | 50 Milligram (mg) Sunitinib
Number analyzed (Participants) | 37
participants | 14

5. Secondary Outcome: Progression-Free Survival (Overall ITT)
Description: Time from start of study treatment to first documentation of objective tumor progression, or to death due to any cause.
Time Frame: From start of treatment until Day 28 of Cycle 1, Day 28 of Cycles thereafter or death
Population: ITT
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | 50 Milligram (mg) Sunitinib
Number analyzed (Participants) | 37
Weeks | 16.1 [8.0 to 28.0]

6. Secondary Outcome: Progression-Free Survival (ITT Child Pugh Class A Subject Population)
Description: Time from start of study treatment to first documentation of objective tumor progression, or to death due to any cause.
Time Frame: From start of treatment until Day 28 of Cycle 1, Day 28 of Cycles thereafter or death
Population: ITT Child Pugh Class A (assessment of liver function) subject population = subjects enrolled in the study with Child-Pugh Class A that received at least 1 dose of study medication.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | 50 Milligram (mg) Sunitinib
Number analyzed (Participants) | 31
Weeks | 21.0 [8.1 to 32.4]

7. Secondary Outcome: Time to Tumor Progression (Overall ITT)
Description: Time from the start of study treatment to the first documentation of objective tumor progression.
Time Frame: From start of treatment until Day 28 of Cycle 1, Day 28 of Cycles thereafter
Population: ITT
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | 50 Milligram (mg) Sunitinib
Number analyzed (Participants) | 37
Weeks | 23.00 [11.71 to 34.14]

8. Primary Outcome: Objective Response (CR or PR)
Description: Number of patients with objective response: confirmed CR or confirmed PR according to RECIST. CR was defined as the disappearance of all target lesions. A PR was defined as a ≥30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions. To be assigned a status of PR or CR, changes in tumor measurements in patients with responding tumors had to have been confirmed by repeat studies that were performed ≥ 4 weeks after the criteria for response were first met.
Time Frame: From start of treatment until Day 28 of Cycle 1, Day 28 of Cycles thereafter
Population: ITT
Measure: Number; unit: participants
Arm/Group | 50 Milligram (mg) Sunitinib
Number analyzed (Participants) | 37
participants | 1
Statistical Analysis 1: Comparison: 50 Milligram (mg) Sunitinib; Test type: Superiority or Other; objective response rate = 2.7, 95% CI [0.1 to 14.2] — percentage of patients with confirmed CR or confirmed PR according to RECIST, relative to the total number of treated patients

9. Secondary Outcome: Time to Tumor Progression (ITT Child Pugh Class A Subject Population)
Description: Time from the start of study treatment to the first documentation of objective tumor progression.
Time Frame: From start of treatment until Day 28 of Cycle 1, Day 28 of Cycles thereafter
Population: ITT Child Pugh Class A (assessment of liver function) subject population
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | 50 Milligram (mg) Sunitinib
Number analyzed (Participants) | 31
Weeks | 23.00 [16.14 to 34.14]

10. Secondary Outcome: Overall Survival (Overall ITT)
Description: Time from the date of first dose of study medication to the date of death due to any cause.
Time Frame: From start of study treatment until death.
Population: ITT
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | 50 Milligram (mg) Sunitinib
Number analyzed (Participants) | 37
Weeks | 34.6 [19.0 to 57.0]

11. Secondary Outcome: Overall Survival (ITT Child Pugh Class A Subject Population)
Description: Time from the date of first dose of study medication to the date of death due to any cause.
Time Frame: From start of study treatment until death.
Population: ITT Child Pugh Class A (assessment of liver function) subject population
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | 50 Milligram (mg) Sunitinib
Number analyzed (Participants) | 31
Weeks | 40.4 [23.4 to 65.1]

12. Secondary Outcome: 1-Year Survival Probability
Description: Probability of survival 1 year after the first dose of study treatment.
Time Frame: From start of treatment until Day 28 of Cycle 1, Day 28 of Cycles thereafter up until 1 year.
Population: ITT
Measure: Number; unit: Probability
Arm/Group | 50 Milligram (mg) Sunitinib
Number analyzed (Participants) | 37
Probability | 0.324
Statistical Analysis 1: Comparison: 50 Milligram (mg) Sunitinib; Test type: Superiority or Other; probability = 0.324, 95% CI [0.168 to 0.479] — probability derived from Kaplan-Meier estimate

13. Secondary Outcome: Trough Plasma Concentrations (Ctrough) of Sunitinib
Description: Ctrough = the concentration prior to study drug administration.
Time Frame: Cycle 1 (Days 1, 14, 28), Cycle 2 (Days 1, 28), Cycle 3 (Days 1, 28), Cycle 5 (Day 28)
Population: Pharmacokinetic (PK) = All subjects enrolled in the study who at least 1 PK sample collected.
Measure: Mean (Standard Deviation); unit: nanograms (ng)/milliliter (mL)
Arm/Group | 50 Milligram (mg) Sunitinib
Number analyzed (Participants) | 37
nanograms (ng)/milliliter (mL)
  Cycle 1, Day 1 (n=37) | 0.00 (0.00)
  Cycle 1, Day 14 (n=32) | 75.05 (35.74)
  Cycle 1, Day 28 (n=29) | 64.19 (38.36)
  Cycle 2, Day 1 (n=25) | 3.27 (6.87)
  Cycle 2, Day 28 (n=19) | 47.68 (39.27)
  Cycle 3, Day 1 (n=16) | 1.11 (1.78)
  Cycle 3, Day 28 (n=16) | 43.92 (26.85)
  Cycle 5, Day 28 (n=12) | 31.99 (18.20)

14. Secondary Outcome: Ctrough of SU-012662 (Metabolite of Sunitinib)
Description: Ctrough = the concentration prior to study drug administration.
Time Frame: Cycle 1 (Days 1, 14, 28), Cycle 2 (Days 1, 28), Cycle 3 (Days 1, 28), Cycle 5 (Day 28)
Population: PK
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 50 Milligram (mg) Sunitinib
Number analyzed (Participants) | 37
ng/mL
  Cycle 1, Day 1 (n=37) | 0.00 (0.00)
  Cycle 1, Day 14 (n=32) | 20.49 (8.68)
  Cycle 1, Day 28 (n=29) | 20.77 (12.93)
  Cycle 2, Day 1 (n=25) | 2.29 (3.55)
  Cycle 2, Day 28 (n=19) | 18.04 (15.02)
  Cycle 3, Day 1 (n=16) | 1.14 (1.48)
  Cycle 3, Day 28 (n=16) | 17.50 (14.20)
  Cycle 5, Day 28 (n=12) | 11.19 (5.81)

15. Secondary Outcome: Ctrough of Total Drug (Sunitinib + SU-012662)
Description: Ctrough = the concentration prior to study drug administration.
Time Frame: Cycle 1 (Days 14, 28), Cycle 2 (Days 1, 28), Cycle 3 (Days 1, 28), Cycle 5 (Day 28)
Population: PK
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 50 Milligram (mg) Sunitinib
Number analyzed (Participants) | 32
ng/mL
  Cycle 1, Day 14 (n=32) | 95.54 (41.72)
  Cycle 1, Day 28 (n=28) | 87.99 (45.21)
  Cycle 2, Day 1 (n=14) | 9.92 (11.52)
  Cycle 2, Day 28 (n=19) | 65.73 (53.39)
  Cycle 3, Day 1 (n=8) | 4.49 (2.98)
  Cycle 3, Day 28 (n=16) | 61.41 (38.95)
  Cycle 5, Day 28 (n=11) | 47.11 (17.84)

16. Secondary Outcome: Dose-Corrected Ctrough of Sunitinib
Description: Data was dose-corrected to the starting dose (dose-corrected Ctrough = observed Ctrough x [starting dose/actual dose]).
Time Frame: Cycle 1 (Days 1, 14, 28), Cycle 2 (Days 1, 28), Cycle 3 (Days 1, 28), Cycle 5 (Day 28)
Population: PK
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 50 Milligram (mg) Sunitinib
Number analyzed (Participants) | 37
ng/mL
  Cycle 1, Day 1 (n=37) | 0.00 (0.00)
  Cycle 1, Day 14 (n=29) | 78.52 (34.97)
  Cycle 1, Day 28 (n=18) | 78.20 (35.44)
  Cycle 2, Day 1 (n=11) | 6.55 (9.08)
  Cycle 2, Day 28 (n=15) | 62.88 (35.27)
  Cycle 3, Day 1 (n=6) | 3.01 (1.67)
  Cycle 3, Day 28 (n=10) | 63.83 (30.77)
  Cycle 5, Day 28 (n=10) | 58.50 (30.39)

17. Secondary Outcome: Dose-Corrected Ctrough of SU-012662 (Metabolite of Sunitinib)
Description: Data was dose-corrected to the starting dose (dose-corrected Ctrough = observed Ctrough x [starting dose/actual dose]).
Time Frame: Cycle 1 (Days 1, 14, 28), Cycle 2 (Days 1, 28), Cycle 3 (Days 1, 28), Cycle 5 (Day 28)
Population: PK
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 50 Milligram (mg) Sunitinib
Number analyzed (Participants) | 37
ng/mL
  Cycle 1, Day 1 (n=37) | 0.00 (0.00)
  Cycle 1, Day 14 (n=29) | 21.07 (8.35)
  Cycle 1, Day 28 (n=18) | 24.20 (10.32)
  Cycle 2, Day 1 (n=12) | 3.63 (2.54)
  Cycle 2, Day 28 (n=15) | 22.86 (14.93)
  Cycle 3, Day 1 (n=7) | 2.71 (1.00)
  Cycle 3, Day 28 (n=10) | 24.67 (17.05)
  Cycle 5, Day 28 (n=10) | 18.38 (8.74)

18. Secondary Outcome: Dose-Corrected Ctrough of Total Drug (Sunitinib + SU-012662)
Description: Data was dose-corrected to the starting dose (dose-corrected Ctrough = observed Ctrough x [starting dose/actual dose]).
Time Frame: Cycle 1 (Days 14, 28), Cycle 2 (Days 1, 28), Cycle 3 (Days 1, 28), Cycle 5 (Day 28)
Population: PK
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 50 Milligram (mg) Sunitinib
Number analyzed (Participants) | 37
ng/mL
  Cycle 1, Day 14 (n=29) | 99.59 (40.43)
  Cycle 1, Day 28 (n=18) | 102.40 (41.92)
  Cycle 2, Day 1 (n=13) | 8.89 (11.08)
  Cycle 2, Day 28 (n=15) | 85.75 (48.87)
  Cycle 3, Day 1 (n=8) | 4.63 (2.85)
  Cycle 3, Day 28 (n=10) | 88.50 (44.20)
  Cycle 5, Day 28 (n=10) | 76.87 (35.89)

19. Secondary Outcome: Circulating Endothelial Cells (CECs) and Circulating Endothelial Progenitor Cells (CEPs)
Description: Blood samples for the assessment of CECs and circulating CEPs were planned to be obtained for subjects in Part 1 of the study, and for a subset of subjects in Part 2 of the study to complete the angiogenic profile of unresectable hepatocellular carcinoma, in addition to the soluble protein evaluation.
Time Frame: Cycle 1 (Days 1, 14), Cycle 2 (Days 1, 28), Cycle 5 (Day 1)
Population: ITT. Blood samples for CECs and CEP cells were collected during the study, but evaluations of these samples were not performed.
Measure: Mean (Standard Deviation); unit: cells/mL
Arm/Group | 50 Milligram (mg) Sunitinib
Number analyzed (Participants) | 0

20. Secondary Outcome: Tissue Tumor Markers Assessed by Tumor Biopsy
Description: Provision of previously collected tumor paraffin blocks (or at least 5-10 4-micron slides prepared from the paraffin block) for correlative laboratory analysis was optional. For all subjects showing OR on study, it was highly recommended to provide previously collected paraffin blocks (or at least 5-10 4-micron slides prepared from the paraffin block). These samples were to be analyzed for markers that may be associated with tumor proliferation or angiogenesis.
Time Frame: Day 28 of Cycle 1 (optional)
Population: ITT. Tumor biopsy results were collected optionally in 5 subjects; however, no evaluations were performed.
Measure: Mean (Standard Deviation); unit: intensity score
Arm/Group | 50 Milligram (mg) Sunitinib
Number analyzed (Participants) | 0

21. Secondary Outcome: Plasma Concentration of Vascular Endothelial Growth Factor (VEGF)
Description: Plasma concentrations of VEGF that may be associated with tumor proliferation or angiogenesis were collected from a subset of subjects and analyzed by e nzyme-linked immunosorbent assay (ELISA). Soluble protein values: Baseline concentration (pM) and ratio to Baseline at each timepoint; ratio to Baseline = plasma concentration of soluble protein at timepoint / concentration of soluble protein at baseline. Samples below the limit of quantitation and samples with insufficient volume available were excluded.
Time Frame: Cycle 1 (Days 1, 14, 28), Cycle 2 (Days 1, 28), Cycle 5 (Day 28)
Population: ITT
Measure: Median (Full Range); unit: picograms (pg)/mL
Arm/Group | 50 Milligram (mg) Sunitinib
Number analyzed (Participants) | 37
picograms (pg)/mL
  Cycle 1, Day 1 (n=37) | 54.9 [20.2 to 466.3]
  Cycle 1, Day 14 (n=33) | 210.7 [71.4 to 2301.8]
  Cycle 1, Day 28 (n=28) | 182.9 [43.6 to 973]
  Cycle 2, Day 1 (n=25) | 81.3 [27.4 to 328.3]
  Cycle 2, Day 28 (n=19) | 234.7 [51.1 to 1717.6]
  Cycle 5, Day 28 (n=12) | 157.8 [91 to 2666.9]

22. Secondary Outcome: Plasma Concentration of VEGF-C
Description: Plasma concentrations of VEGF-C that may be associated with tumor proliferation or angiogenesis were collected from a subset of subjects and analyzed by ELISA. Soluble protein values: Baseline concentration (pM) and ratio to Baseline at each timepoint; ratio to Baseline = plasma concentration of soluble protein at timepoint / concentration of soluble protein at baseline. Samples below the limit of quantitation and samples with insufficient volume available were excluded.
Time Frame: Cycle 1 (Days 1, 14, 28), Cycle 2 (Days 1, 28), Cycle 5 (Day 28)
Population: ITT
Measure: Median (Full Range); unit: pg/mL
Arm/Group | 50 Milligram (mg) Sunitinib
Number analyzed (Participants) | 37
pg/mL
  Cycle 1, Day 1 (n=37) | 822.2 [334.5 to 3216.5]
  Cycle 1, Day 14 (n=33) | 731.7 [394.6 to 3540.5]
  Cycle 1, Day 28 (n=28) | 693.1 [336.4 to 1862.3]
  Cycle 2, Day 1 (n=25) | 733.8 [457.9 to 1390.3]
  Cycle 2, Day 28 (n=19) | 601.6 [339.9 to 1565.4]
  Cycle 5, Day 28 (n=12) | 802.7 [441.9 to 2268.7]

23. Secondary Outcome: Plasma Concentration of Soluble VEGF Receptor-2 (sVEGFR-2)
Description: Plasma concentrations of sVEGFR-2 that may be associated with tumor proliferation or angiogenesis were collected from a subset of subjects and analyzed by ELISA. Soluble protein values: Baseline concentration (pM) and ratio to Baseline at each timepoint; ratio to Baseline = plasma concentration of soluble protein at timepoint / concentration of soluble protein at baseline). Samples below the limit of quantitation and samples with insufficient volume available were excluded.
Time Frame: Cycle 1 (Days 1, 14, 28), Cycle 2 (Days 1, 28), Cycle 5 (Day 28)
Population: ITT
Measure: Median (Full Range); unit: pg/mL
Arm/Group | 50 Milligram (mg) Sunitinib
Number analyzed (Participants) | 37
pg/mL
  Cycle 1, Day 1 (n=37) | 7068.5 [4572.5 to 13667.5]
  Cycle 1, Day 14 (n=33) | 3824.5 [2044.5 to 9404]
  Cycle 1, Day 28 (n=28) | 3105.8 [1566 to 9391.5]
  Cycle 2, Day 1 (n=25) | 6121.5 [2604 to 12471]
  Cycle 2, Day 28 (n=19) | 3542 [2148 to 9416.5]
  Cycle 5, Day 28 (n=12) | 4408.5 [1742 to 10612]

24. Secondary Outcome: Plasma Concentration of Soluble VEGF Receptor-3 (sVEGFR-3)
Description: Plasma concentrations of sVEGFR-3 that may be associated with tumor proliferation or angiogenesis were collected from a subset of subjects and analyzed by ELISA. Soluble protein values: Baseline concentration (pM) and ratio to Baseline at each timepoint; ratio to Baseline = plasma concentration of soluble protein at timepoint / concentration of soluble protein at baseline. Samples below the limit of quantitation and samples with insufficient volume available were excluded.
Time Frame: Cycle 1 (Days 1, 14, 28), Cycle 2 (Days 1, 28), Cycle 5 (Day 28)
Population: ITT
Measure: Median (Full Range); unit: pg/mL
Arm/Group | 50 Milligram (mg) Sunitinib
Number analyzed (Participants) | 37
pg/mL
  Cycle 1, Day 1 (n=37) | 48700 [12420 to 119300]
  Cycle 1, Day 14 (n=33) | 25300 [5760 to 79000]
  Cycle 1, Day 28 (n=28) | 11075 [3060 to 54050]
  Cycle 2, Day 1 (n=25) | 44100 [6820 to 95900]
  Cycle 2, Day 28 (n=19) | 11450 [4920 to 44870]
  Cycle 5, Day 28 (n=12) | 12430 [6230 to 72300]

25. Secondary Outcome: Plasma Concentration of Soluble KIT (sKIT)
Description: Plasma concentrations of sKIT that may be associated with tumor proliferation or angiogenesis were collected from a subset of subjects and analyzed by ELISA analysis. Soluble protein values: Baseline concentration (pM) and ratio to Baseline at each timepoint; ratio to Baseline = plasma concentration of soluble protein at timepoint / concentration of soluble protein at baseline. Samples below the limit of quantitation and samples with insufficient volume available were excluded.
Time Frame: Cycle 1 (Days 1, 14, 28), Cycle 2 (Days 1, 28), Cycle 5 (Day 28)
Population: ITT
Measure: Median (Full Range); unit: pg/mL
Arm/Group | 50 Milligram (mg) Sunitinib
Number analyzed (Participants) | 37
pg/mL
  Cycle 1, Day 1 (n=37) | 41960 [17560 to 85345]
  Cycle 1, Day 14 (n=33) | 32680 [14005 to 57840]
  Cycle 1, Day 28 (n=28) | 22910 [12710 to 37400]
  Cycle 2, Day 1 (n=25) | 21615 [9520 to 41855]
  Cycle 2, Day 28 (n=19) | 18125 [10995 to 35940]
  Cycle 5, Day 28 (n=12) | 18420 [8265 to 29115]

ADVERSE EVENTS:
Arm/Group | 50 Milligram (mg) Sunitinib
Serious Adverse Events (participants affected / at risk) | 24/37
Other Adverse Events (participants affected / at risk) | 37/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 50 Milligram (mg) Sunitinib (N=37)
Anaemia (Blood and lymphatic system disorders) | 6
Leukopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 6
Myocardial infarction (Cardiac disorders) | 1
Cataract (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3
Gingival bleeding (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 2
Mouth haemorrhage (Gastrointestinal disorders) | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 4
Peritoneal effusion (Gastrointestinal disorders) | 1
Peritoneal haemorrhage (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 2
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 5
Hypothermia (General disorders) | 1
Pain (General disorders) | 1
Pyrexia (General disorders) | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Empyema (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Aphasia (Nervous system disorders) | 1
Balance disorder (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Coma (Nervous system disorders) | 1
Depressed level of consciousness (Nervous system disorders) | 1
Hepatic encephalopathy (Nervous system disorders) | 3
Loss of consciousness (Nervous system disorders) | 1
Nervous system disorder (Nervous system disorders) | 1
Neurological decompensation (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 4
Confusional state (Psychiatric disorders) | 2
Renal failure (Renal and urinary disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 50 Milligram (mg) Sunitinib (N=37)
Anaemia (Blood and lymphatic system disorders) | 9
Leukopenia (Blood and lymphatic system disorders) | 7
Neutropenia (Blood and lymphatic system disorders) | 8
Thrombocytopenia (Blood and lymphatic system disorders) | 17
Vertigo (Ear and labyrinth disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 8
Abdominal pain upper (Gastrointestinal disorders) | 8
Ascites (Gastrointestinal disorders) | 9
Constipation (Gastrointestinal disorders) | 7
Diarrhoea (Gastrointestinal disorders) | 16
Dry mouth (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 7
Dysphagia (Gastrointestinal disorders) | 5
Gastritis (Gastrointestinal disorders) | 2
Gingivitis (Gastrointestinal disorders) | 2
Haematemesis (Gastrointestinal disorders) | 2
Haemorrhoids (Gastrointestinal disorders) | 2
Melaena (Gastrointestinal disorders) | 2
Mouth haemorrhage (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 17
Odynophagia (Gastrointestinal disorders) | 2
Stomatitis (Gastrointestinal disorders) | 9
Varices oesophageal (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 9
Asthenia (General disorders) | 17
Chest pain (General disorders) | 2
Face oedema (General disorders) | 4
Fatigue (General disorders) | 5
Malaise (General disorders) | 4
Mucosal inflammation (General disorders) | 7
Oedema peripheral (General disorders) | 6
Pain (General disorders) | 2
Pitting oedema (General disorders) | 3
Pyrexia (General disorders) | 7
Hepatic pain (Hepatobiliary disorders) | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 6
Bronchitis (Infections and infestations) | 2
Fungal skin infection (Infections and infestations) | 3
Skin infection (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 3
Fall (Injury, poisoning and procedural complications) | 2
Alanine aminotransferase increased (Investigations) | 6
Aspartate aminotransferase increased (Investigations) | 7
Blood alkaline phosphatase increased (Investigations) | 3
Blood bilirubin (Investigations) | 2
Gamma-glutamyltransferase increased (Investigations) | 5
Haemoglobin (Investigations) | 3
Platelet count (Investigations) | 3
Weight decreased (Investigations) | 6
White blood cell count (Investigations) | 4
Anorexia (Metabolism and nutrition disorders) | 17
Dehydration (Metabolism and nutrition disorders) | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 4
Hypoglycaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 3
Hyponatraemia (Metabolism and nutrition disorders) | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Ageusia (Nervous system disorders) | 3
Dizziness (Nervous system disorders) | 2
Dysgeusia (Nervous system disorders) | 4
Headache (Nervous system disorders) | 8
Neuropathy peripheral (Nervous system disorders) | 2
Sciatica (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 2
Confusional state (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 7
Erythema (Skin and subcutaneous tissue disorders) | 2
Hair colour changes (Skin and subcutaneous tissue disorders) | 6
Nail disorder (Skin and subcutaneous tissue disorders) | 2
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 11
Periorbital oedema (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 5
Skin discolouration (Skin and subcutaneous tissue disorders) | 6
Skin exfoliation (Skin and subcutaneous tissue disorders) | 2
Skin irritation (Skin and subcutaneous tissue disorders) | 3
Skin lesion (Skin and subcutaneous tissue disorders) | 4
Hypertension (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of <60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), <12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential info other than study results.